CLINICAL TRIAL: NCT07135648
Title: A Single-center, Randomized, Controlled, Partially Blinded, Crossover Study to Evaluate the Nicotine Pharmacokinetics and Pharmacodynamics of Two Variants of Vibrating Mesh 1.0 (VM 1.0), a Nicotine-containing Aerosol Generator, Compared to Cigarettes in Adult Current Smokers
Brief Title: Nicotine Pharmacokinetics and Pharmacodynamics of Two Variants of VM 1.0 Compared to Cigarettes in Adult Current Smokers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Philip Morris Products S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: NS-VM-PK-01
Record Dates: First submitted 2025-08-14; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Nicotine
MeSH Terms: interventions — Tobacco Products

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This is a partially blinded study: the participants will be blinded to the variants of VM 1.0 and to the randomized product use sequences. As part of the PMP quality control (QC) activity, a blinded data review will be performed before database lock. Data listings will be reviewed by the CRO and PMP, with no access to the product information for data review team members. Full details will be available in the data review plan.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Product Sequence 1 (Active Comparator): On Day 1 to Day 3, after at least 10 hours of abstinence from any nicotine/tobacco containing products and after at least 10 hours of fasting, participants will use one of the three investigational products according to randomized product use sequence and as instructed by the investigational site personnel.
  The list of possible sequences are:
  Cigarette; VM32; VM16 / VM16; Cigarette; VM32 / VM32; VM16; Cigarette
  Interventions: Other: VM16; Other: VM32; Other: Cigarette (CC)
- Product Sequence 2 (Active Comparator): On Day 1 to Day 3, after at least 10 hours of abstinence from any nicotine/tobacco containing products and after at least 10 hours of fasting, participants will use one of the three investigational products according to randomized product use sequence and as instructed by the investigational site personnel.
  The list of possible sequences are:
  Cigarette; VM32; VM16 / VM16; Cigarette; VM32 / VM32; VM16; Cigarette
  Interventions: Other: VM16; Other: VM32; Other: Cigarette (CC)
- Product Sequence 3 (Active Comparator): On Day 1 to Day 3, after at least 10 hours of abstinence from any nicotine/tobacco containing products and after at least 10 hours of fasting, participants will use one of the three investigational products according to randomized product use sequence and as instructed by the investigational site personnel.
  The list of possible sequences are:
  Cigarette; VM32; VM16 / VM16; Cigarette; VM32 / VM32; VM16; Cigarette
  Interventions: Other: VM16; Other: VM32; Other: Cigarette (CC)

INTERVENTIONS:
Other: VM16 — VM16 contains a liquid with a nicotine concentration of 1.6%
Other: VM32 — VM32 contains a liquid with a nicotine concentration of 3.2%
Other: Cigarette (CC) — Subjects will provide their own usual brand of commercially available cigarettes

SUMMARY:
A single-center, randomized, controlled, partially blinded, crossover study to evaluate the pharmacokinetics and pharmacodynamics of nicotine following use of two variants of VM 1.0, VM16 and VM32, a nicotine-containing aerosol generator compared to cigarettes in adult current smokers. The participants will be blinded to the variants of VM 1.0 and to the randomized product use sequences. The study will be conducted with 3 periods and 3 sequences.

ELIGIBILITY:
Inclusion Criteria:

* Participant has signed the ICF and is able to understand the information provided in the ICF.
* Male or female participant between 21 and 65 years inclusive.
* Participant has smoked commercially available or roll-your own cigarettes (no brand restrictions) for at least the last 12 months prior to the Screening visit.
* Participant has smoked at least 10 commercially available cigarettes per day in the past 30 days prior to the Screening visit and Admission.
* Nicotine exposure status will be verified by urinary cotinine test (cotinine ≥ 200 ng/mL).
* Participant has a BMI >18.5 and <30.0 kg/m2 and body weight ≥50.0 kg for males and ≥45.0 kg for females.
* Participant is available for the entire study period and willing to comply with study procedures, including product use assignments and periods of abstinence from any nicotine/tobacco containing products and willing to adhere to a standardized diet.

Exclusion Criteria:

* Participant has reasons other than medical (e.g., psychological, social reason) not to be part of the study, as determined by the Principal Investigator or designee.
* Participant is legally incompetent, or physically or mentally incapable of giving consent (e.g., emergency situation, under guardianship, prisoners).
* Participant has a health condition which requires medication or any other clinically significant finding e.g., safety labs, pulmonary function test, vital signs, physical examination, ECG and medical history, as determined by the Principal Investigator or designee.
* Participant experiences difficulty with venipuncture and/or poor venous access.
* Participant has medical conditions which require, or will require during the study, a medical intervention (e.g., start of treatment, surgery, hospitalization).
* Presence of fever (body temperature >37.5°C) e.g., a fever associated with a symptomatic viral or bacterial infection.
* Participant has a hemoglobin level < 11.0 g/dL for females and < 12.0 g/dL for males at the Screening visit.
* Participant uses medication that aids in smoking cessation.
* Participant uses Tetrahydrocannabinol (THC)-containing products.
* Participant previously attempted to quit using tobacco- or nicotine-containing products within 28 days prior to Admission.
* Participant has donated plasma within seven days prior to screening or has donated or lost 450 mL or more of whole blood within 8 weeks prior to Screening for males, and in the 12 weeks prior to the Screening visit for females.
* Participant has a positive serology test for HIV 1/2, hepatitis B or C.
* Participant has a medical history of alcohol abuse within one year prior to Screening or regular use of alcohol within six months prior to the Screening visit that exceeds 10 units for women or 15 units for men of alcohol per week.
* Participant has a positive urine drug test.
* Participant has a positive alcohol breath test.
* Participant or one of their family members is a current or former employee of the tobacco industry.
* Participant or one of their family members is an employee of the investigational site or of any other parties involved in the study.
* Participant has participated in another clinical study within 30 days prior to the Screening visit or concomitantly participates in any other investigational study.
* Participant has been previously screened or enrolled in this study (except alternates)
* For female participants only: participant has a positive urine pregnancy test at the Screening visit or at Admission or is a breastfeeding.
* For females of childbearing potential only: participant does not agree to use an acceptable method of effective contraception.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2025-07-17 (Actual); Primary Completion 2025-07-28 (Actual); Study Completion 2025-10-06 (Estimated)

PRIMARY OUTCOMES:
Nicotine concentration | From 5 minutes prior to product use to 12 hours after product use
  To measure the observed plasma nicotine concentration [C -5min] and [C 12hours], to describe the plasma concentration-time profile of nicotine and derived pharmacokinetic (PK) parameters from VM16 and VM32 use with a fixed puffing regimen and single cigarette smoking.
Maximum nicotine concentration | From 5 minutes prior to product use to 12 hours after product use
  To measure the maximum observed plasma nicotine concentration [Cmax], to describe the plasma concentration-time profile of nicotine and derived pharmacokinetic (PK) parameters from VM16 and VM32 use with a fixed puffing regimen and single cigarette smoking.
Area under the observed plasma nicotine concentration-time curve (AUC) | From 5 minutes prior to product use to 12 hours after product use
  To measure the area under the observed plasma nicotine concentration-time curve (AUC) from the start the first puff (T0) to the timepoint of last quantifiable concentration [AUC 0-last] and extrapolated to infinity [AUC 0-infinity]
Time to the observed maximum concentration [Tmax] | From 5 minutes prior to product use to 12 hours after product use
  To measure the time to the observed maximum concentration [Tmax], to describe the plasma concentration-time profile of nicotine and derived pharmacokinetic (PK) parameters from VM16 and VM32 use with a fixed puffing regimen and single cigarette smoking.
Elimination rate constant [kel] | From 5 minutes prior to product use to 12 hours after product use
  To measure the elimination rate constant [kel]], to describe the plasma concentration-time profile of nicotine and derived pharmacokinetic (PK) parameters from VM16 and VM32 use with a fixed puffing regimen and single cigarette smoking.
Half-life of nicotine [t1/2] | From 5 minutes prior to product use to 12 hours after product use
  To measure half-life of nicotine [t1/2], to describe the plasma concentration-time profile of nicotine and derived pharmacokinetic (PK) parameters from VM16 and VM32 use with a fixed puffing regimen and single cigarette smoking.

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Jaumont, MD, Study Chair — Philip Morris Products S.A.
Locations (1):
- Celerion, Belfast, United Kingdom

IPD SHARING:
Plan to Share IPD: No